CLINICAL TRIAL: NCT01606215
Title: Stem Cells in Rapidly Evolving Active Multiple Sclerosis
Acronym: STREAMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO1959; 13HH0228 (Other: Imperial College)
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; mesenchymal stem cells; bone marrow; rapidly evolving
MeSH Terms: conditions — Multiple Sclerosis | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental): 1-2 x106 MSCs/kg administered at Week 0
  Interventions: Drug: Mesenchymal stem cells
- Placebo (Sham Comparator): Suspension media administered at Week 0
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesenchymal stem cells — 1.0-2.0 million cells/kg body weight
  Other Names: Mesenchymal stromal cells
  Arms: mesenchymal stem cells
Drug: Placebo — Placebo
  Other Names: Sham
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind crossover study to study the effect of intravenous treatment with autologous (derived from the individuals themselves) mesenchymal stem cells (MSCs) in patients with multiple sclerosis (MS).

DETAILED DESCRIPTION:
Current treatments for MS target the immune system and are not curative. There is much interest in MSCs as they have the potential to not only affect the immune system but may also promote repair. This study will use MSCs that are harvested from the bone marrow and grown for up to 52 days before being given back to the person from whom they were harvested. This avoids any chemotherapy so is therefore safer than other types of stem cells. In this crossover study, everyone will receive their own stem cells back but in half of the patients it will be delayed by 24 weeks.

The primary outcomes are to check that the procedure is safe and to measure any changes on the MRI at 24 weeks. Other more exploratory measures will try to assess effects on repair in the central nervous system (CNS).

ELIGIBILITY:
Inclusion Criteria:

Patients with clinically and radiologically active multiple sclerosis as defined by:

1. Diagnosis of MS:

   * Relapsing remitting MS (RRMS): ≥ 1 moderate-severe relapse and ≥1 GEL in past 18 months or ≥ 1 moderate-severe relapse and ≥1 new T2 lesion in past 18 months.
   * Secondary progressive MS (SPMS) with an increase of ≥ 1 EDSS point (if baseline EDSS ≤ 5) or 0.5 EDSS point (if baseline EDSS ≥ 5.5), in the previous 18 months and ≥ 1 GEL in past 18 months or ≥ 1 moderate-severe relapse and ≥1 new T2 lesion in past 18 months.
   * Primary progressive MS (PPMS) patients with positive oligoclonal bands (OCBs) in the cerebrospinal fluid (CSF) and an increase of ≥ 1 EDSS point (if baseline EDSS is ≤ 5.0) or 0.5 EDSS point (if baseline EDSS is ≥ 5.5), or quantifiable, objective evidence of equivalent progression in the previous 18 months and ≥ 1 GEL in past 18 months or ≥ 1 new T2 lesion in past 18 months.
2. Age 18 to 50 years.
3. Disease duration 2 to 10 years from diagnosis (inclusive).
4. Expanded Disability Status Scale (EDSS) 2.0 to 6.5 at screening evaluation.
5. ≥ 1 GEL on MRI within 6 months prior to harvesting.
6. Adequate culture of a subject's MSCs and their release for clinical use.

Exclusion Criteria:

1. RRMS without at least one severe relapse in the previous 18 months or without at least one GEL or one new T2 in the previous 18 months.
2. SPMS without relapses and without new lesions (GEL or T2 positive) at MRI in the last 18 months.
3. PPMS without positive CSF OCBs or without a GEL or new T2 lesion in the previous 18 months.
4. No gadolinium enhancing lesion(s) in the 3 months prior to bone marrow harvesting.
5. A previously ineligible patient who failed to meet the MRI requirements of the inclusion criteria will not be reviewed again even if further imaging, revealing ≥ 1 GEL, becomes available.
6. Failure of bone marrow (BM) sample to generate MSCs suitable for clinical use within a specified time frame (4 weeks).
7. Treatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the last 3 months.
8. Treatment with interferon-beta or glatiramer acetate within the last 1 month.
9. Treatment with alemtuzumab (campath-1H) within the last 2 years.
10. Prior treatment with total lymphoid irradiation and autologous or allogeneic hematopoietic stem cell transplantation.
11. Participation in clinical trials of any experimental drugs in the 6 months before study entry.
12. Corticosteroid treatment in the last 30 days.
13. Presence of any active or chronic infection.
14. Previous history of a malignancy other than basal cell carcinoma of the skin and carcinoma in situ that has been in remission for more than one year.
15. Severely limited life expectancy by any other co-morbid illness.
16. Abnormal blood counts, a history of myelodysplasia or other cytopenia.
17. Known pregnancy, positive urine pregnancy test at screening or risk or pregnancy (this includes patients who are unwilling to practice active contraception during the duration of the study).
18. Contraindication to MRI including but not limited to intracranial aneurysm clips (except Sugita), history of intra-orbital metal fragments that have not been removed by an MD (as confirmed by orbital X-Ray), pacemaker and non-MRI compatible devices (e.g. heart valves, inner ear implants), history of claustrophobia or the inability of the subject to lie still on their back for a period of 1.5 hours in the MRI scanner.
19. An estimated glomerular filtration rate (eGFR)< 60 mL/min/1.73m2 or history or presence of renal impairment (e.g. serum creatinine clearance less than 30ml/min).
20. Inability to give written informed consent/comply with study procedures.
21. Any significant organ dysfunction or co-morbidity that the Investigators consider would put the subject at unacceptable risk by participating in the study or that would interfere with the functional assessments.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo A Muraro, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uccelli A, Laroni A, Brundin L, Clanet M, Fernandez O, Nabavi SM, Muraro PA, Oliveri RS, Radue EW, Sellner J, Soelberg Sorensen P, Sormani MP, Wuerfel JT, Battaglia MA, Freedman MS; MESEMS study group. MEsenchymal StEm cells for Multiple Sclerosis (MESEMS): a randomized, double blind, cross-over phase I/II clinical trial with autologous mesenchymal stem cells for the therapy of multiple sclerosis. Trials. 2019 May 9;20(1):263. doi: 10.1186/s13063-019-3346-z. PMID 31072380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 patients screened into trial and having bone marrow aspiration
Pre-assignment Details: Bone marrow aspiration and expansion in the stem cell laboratory. Continuation in trial required expansion of MSCs to 1-2 x106 million MSCs/kg Of the 21 patients screened, only 13 continued in the trial (others failed MSC expansion and do not contribute to results)
Groups:
- A: Mesenchymal Stem Cells First, Then Placebo: 1-2 x106 MSCs/kg administered at Week 0
  Mesenchymal stem cells: 1.0-2.0 million cells/kg body weight
- B: Placebo First, Then MSCs: Suspension media administered at Week 0
  Placebo: Placebo
Period: Treatment to 1st Group - Placebo to 2nd
Arm/Group | A: Mesenchymal Stem Cells First, Then Placebo | B: Placebo First, Then MSCs
Started | 10 | 11
Completed | 6 | 7
Not Completed | 4 | 4
Not completed — Failure to expand autologous mesenchymal stem cell product according to protocol specifications | 4 | 4
Period: Follow-up
Arm/Group | A: Mesenchymal Stem Cells First, Then Placebo | B: Placebo First, Then MSCs
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Placebo to 1st Group - Treatment to 2nd
Arm/Group | A: Mesenchymal Stem Cells First, Then Placebo | B: Placebo First, Then MSCs
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients for whom MSCs were successfully expanded after the bone marrow aspirate
Groups:
- A: Mesenchymal Stem Cells First, Then Placebo: Mesenchymal stem cells first, then placebo:
  Mesenchymal stem cells; 1.0-2.0 million cells/kg body weight (1-2 x106 MSCs/kg administered at Week 0)
- B: Placebo First, Then MSCs: Placebo first, then MSCs:
  Placebo; Placebo (Suspension media administered at Week 0)
- Total: Total of all reporting groups
Arm/Group | A: Mesenchymal Stem Cells First, Then Placebo | B: Placebo First, Then MSCs | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race | 6 | 7 | 13
  Ethnicity | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Assessed by CTCAE v4.0
Description: The number of adverse events before crossover in the stem cell treatment group compared to the placebo group over the first 24 weeks (please refer to period 1 of the participant flow).
Time Frame: 24 weeks from baseline
Measure: Number; unit: total events
Arm/Group | A: Mesenchymal Stem Cells First, Then Placebo | B: Placebo First, Then MSCs
Number analyzed (Participants) | 6 | 7
total events | 5 | 0

2. Primary Outcome: Number of GELs Newly Appearing at Weeks 4, 12 and 24 After MSC Therapy in the First 24 Weeks of Trial
Description: Where GELs stands for gadolinium enhancing lesions and MSC for Mesenchymal Stem Cell.
  This was to evaluate the efficacy of autologous mesenchymal stem cells in MS patients, quantified by the reduction in the number of new gadolinium-enhancing lesions counted on MRI scans over 24 weeks and the total number of GELs counted over months 1, 3 and 6 will be compared between treatment groups.
Time Frame: Up to 24 weeks
Population: Comparison of GELs between MSC- vs placebo- treated groups up to Week 24
Measure: Mean (Standard Deviation); unit: number of GELS counted
Groups:
- A: Mesenchymal Stem Cells First Then Placebo: 1-2 x106 MSCs/kg administered at Week 0
  Mesenchymal stem cells: 1.0-2.0 million cells/kg body weight
Arm/Group | A: Mesenchymal Stem Cells First Then Placebo | B: Placebo First, Then MSCs
Number analyzed (Participants) | 6 | 7
number of GELS counted
  Week 0 to 4 | 1.5 (2.07) | 1.29 (2.98)
  Week 4 to 12 | 1.5 (2.25) | 2.29 (4.39)
  Week 12 to 24 | 1.17 (0.75) | 2.43 (4.89)
Statistical Analysis 1: Comparison: A: Mesenchymal Stem Cells First Then Placebo vs B: Placebo First, Then MSCs; Week 4 data; Test type: Other; p = 0.84, t-test, 2 sided
Statistical Analysis 2: Comparison: A: Mesenchymal Stem Cells First Then Placebo vs B: Placebo First, Then MSCs; Week 12 data; Test type: Other; p = 0.62, t-test, 2 sided
Statistical Analysis 3: Comparison: A: Mesenchymal Stem Cells First Then Placebo vs B: Placebo First, Then MSCs; Week 24 data; Test type: Other; p = 0.61, t-test, 2 sided

3. Secondary Outcome: Number of Newly Appearing GELs Over Months 1, 3 and 6 Will be Compared Between Treatment Groups.
Description: Number of gadolinium enhancing lesions identified over months 1, 3 and 6 will be compared between treatment groups - the treatment groups in this section relate to all 13 patients treated with MSCs (so patients in arm MSCs first, then placebo and 7 patients in placebo first, then MSCs) with 7 placebo patients (placebo first, then MSCs - the placebo group here ignores the 6 pts treated with MSCs first as we do not know whether there is any ongoing effect of MSCs beyond 24 weeks).
Time Frame: Months 1, 3 and 6
Measure: Mean (Standard Deviation); unit: number of GELS counted
Groups:
- A/B: All Patients Treated With Mesenchymal Stem Cells: 1-2 x106 MSCs/kg administered at Week 0 or Week 24
  Mesenchymal stem cells: 1.0-2.0 million cells/kg body weight
- A: Placebo: Suspension media administered at Week 0
  Placebo: Placebo
Arm/Group | A/B: All Patients Treated With Mesenchymal Stem Cells | A: Placebo
Number analyzed (Participants) | 13 | 7
number of GELS counted
  Week 0 to 4 | 1.38 (1.71) | 1.29 (2.98)
  Week 4 to 12 | 1.92 (2.75) | 2.29 (4.39)
  Week 12 to 24 | 1.46 (1.90) | 2.43 (4.89)

4. Secondary Outcome: Comparison of Contrast Enhancing Lesions Between Treatment Periods Following Crossover
Description: The number of contrast enhancing lesions counted over months 7, 9 and 12 (that is after cross-over).
Time Frame: Months 6-12
Population: crossover phase of trial; weeks 24-48
Measure: Mean (Standard Deviation); unit: number of GELS counted
Groups:
- A: Mesenchymal Stem Cells First, Then Placebo: 1-2 x106 MSCs/kg administered at Week 0; received placebo at Week 24
  Mesenchymal stem cells: 1.0-2.0 million cells/kg body weight
- B: Placebo First, Then MSCs: Suspension media administered at Week 0; received 1-2 x 106MSCs/kg at Week 24
  Placebo: Placebo
Arm/Group | A: Mesenchymal Stem Cells First, Then Placebo | B: Placebo First, Then MSCs
Number analyzed (Participants) | 6 | 7
number of GELS counted
  Week 28 | 2.5 (2.35) | 1.29 (1.50)
  Week 36 | 2.33 (2.94) | 2.29 (3.25)
  Week 48 | 1.5 (1.87) | 1.71 (2.56)

5. Secondary Outcome: Combined Unique MRI Activity
Description: To evaluate the efficacy of autologous mesenchymal stem cells in MS patients, quantified by the reduction in combined unique MRI activity on MRI scans over 24 weeks. The total number of such lesions counted over Weeks 4, 12 and 24 will be compared between treatment groups.
  Combined Unique MRI activity defined as number of new T1w contrast-enhanced lesions plus number of new T2w lesions without contrast enhancement on T1w plus number of enlarging T2w lesions (>50% volume increase, no lesion fusion) without contrast enhancement on T1w.
Time Frame: Weeks 4, 12 and 24
Population: after crossover treatment
Measure: Mean (Standard Deviation); unit: combined unique MRI activity
Groups:
- A: Mesenchymal Stem Cells: 1-2 x106 MSCs/kg first
  Mesenchymal stem cells: 1.0-2.0 million cells/kg body weight second
- B: Placebo: Suspension media first
  Placebo: Placebo second
Arm/Group | A: Mesenchymal Stem Cells | B: Placebo
Number analyzed (Participants) | 6 | 7
combined unique MRI activity
  Week 4 | 1.5 (2.07) | 2 (3.70)
  Week 12 | 2.17 (3.07) | 3.14 (5.05)
  Week 24 | 1.83 (1.60) | 4.43 (8.90)
Statistical Analysis 1: Comparison: A: Mesenchymal Stem Cells vs B: Placebo; Week 4; Test type: Other; p = 0.77, t-test, 2 sided
Statistical Analysis 2: Comparison: A: Mesenchymal Stem Cells vs B: Placebo; Week 12; Test type: Other; p = 0.68, t-test, 2 sided
Statistical Analysis 3: Comparison: A: Mesenchymal Stem Cells vs B: Placebo; Week 24; Test type: Other — Week 24; p = 0.48, t-test, 2 sided

6. Secondary Outcome: Relapses
Description: number of relapses in MSC treatment group vs. placebo group in the first 6 months
Time Frame: 6 months
Measure: Number; unit: total events
Groups:
- A: Mesenchymal Stem Cells: 1-2 x106 MSCs/kg administered at Week 0
  Mesenchymal stem cells: 1.0-2.0 million cells/kg body weight
- B: Placebo: Suspension media administered at Week 0
  Placebo: Placebo
Arm/Group | A: Mesenchymal Stem Cells | B: Placebo
Number analyzed (Participants) | 6 | 7
total events | 2 | 10

7. Secondary Outcome: Progression of Disability
Description: EDSS at 6 months in both groups at Week 24: comparing 'MSCs first, then placebo' and 'Placebo first, then MSCs' at Week 24.
  EDSS is a disability score. EDSS is an abbreviation for Expanded Disability Status Scale. Ranges from 0 (no disability) to 10 (death). A higher score indicates worsening disability.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale (EDSS)
Arm/Group | A: Mesenchymal Stem Cells First, Then Placebo | B: Placebo First, Then MSCs
Number analyzed (Participants) | 6 | 7
score on a scale (EDSS) | 4.0 (1.0) | 3.9 (1.77)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- A: Mesenchymal Stem Cell Tratment First: 1-2 x106 MSCs/kg administered first
  Mesenchymal stem cells: 1.0-2.0 million cells/kg body weight second
- B: Placebo First: Suspension media administered first
  Placebo: Placebo second
Arm/Group | A: Mesenchymal Stem Cell Tratment First | B: Placebo First
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 5/10 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Mesenchymal Stem Cell Tratment First (N=10) | B: Placebo First (N=11)
tinnitus (Ear and labyrinth disorders) | 1 (1) | NA
back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | NA
urinary tract infection (Renal and urinary disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-12-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT01606215/Prot_SAP_ICF_000.pdf